CLINICAL TRIAL: NCT01514760
Title: A Pilot and Feasibility Study of Mobile-Based Asthma Action Plans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 133343
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Adolescents; Mobile based applications; Asthma action plan; Self Efficacy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mobile-based Asthma Action Plan (Experimental): The mobile phone based application features will include ambulatory peak flow and asthma symptoms diary, individualized treatment plan for routine care and during episodes of acute asthma symptoms, and education components to reinforce asthma self-management concepts.
  Interventions: Other: Mobile-based Asthma Action Plan

INTERVENTIONS:
Other: Mobile-based Asthma Action Plan — The participant will be distributed a mobile phone (iPhone or Android) at the time of consent. The mobile-based Asthma Action Plan application will be provided on the mobile device. The mobile phone based application features will include ambulatory peak flow and asthma symptoms diary, individualized treatment plan for routine care and during episodes of acute asthma symptoms, and education components to reinforce asthma self-management concepts. Participants will receive 3 daily messages from the Asthma Action Plan mobile application. A fourth "rotating" message will be sent twice weekly.

SUMMARY:
Investigators from University of Arkansas for Medical Sciences Department of Pediatrics and University of Arkansas for Medical Sciences Center for Distance Health will collaborate to develop a mobile-based Asthma Action Plan application to improve asthma self-management skills specifically targeting adolescents. The investigators hypothesize that an interactive, mobile-based asthma action plan will be a feasible means of reinforcing long-term asthma management guidelines as well as delivering acute management instructions to adolescents with asthma.

DETAILED DESCRIPTION:
A written Asthma Action Plan from a healthcare provider is one of the key features of asthma self-management recommended by the National Asthma Education and Prevention Program asthma guidelines; guidelines-based asthma care has not yet fully translated to the community despite the fact that National Asthma Education and Prevention Program released the first set of national guidelines nearly 2 decades ago. Previous reports have proven that patients with an Asthma Action Plan have better outcomes including fewer acute healthcare utilization visits, fewer days missed from school, and improved symptoms scores compared to patients without an Asthma Action Plan. Recently, mobile-based phone applications and music file (MPEG layer 3)(MP3) players have been utilized in the management of chronic diseases such as asthma and diabetes to provide medication reminders and to provide alternatives to paper dairies for logging symptoms or other health-related data such as peak flow readings or blood glucose readings. We propose to design an application that will fully meet the recommended individualized Asthma Action Plan treatment plan as recommended by national guidelines and will also provide participants with medication reminders, education tips, and data logging/tracking capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 and ≤ 17 years.
* Mild to severe persistent asthma or poorly controlled asthma. If a child has used a preventive medication in the past, but reports no use of the medication in the prior 3 months, we will assess severity.
* Children not using a preventive medication at baseline: We will assess for mild persistent to severe persistent asthma. Any one of the following, during the prior 4 weeks (as defined by parent interview) will determine severity:
* An average of >2 days per week with asthma symptoms
* >2 days per week with rescue medication use
* ≥2 nights per month awakened with nighttime symptoms
* Minor limitation of activity
* ≥2 episodes of asthma during the past year that have required systemic corticosteroids.
* Children using a preventive medication at baseline: We will assess for poorly controlled asthma. Any 1 of the following, during the prior 4 weeks (as defined by parent interview in the waiting room) will determine control:
* An average of >2 days per week with asthma symptoms
* >2 days per week with rescue medication use
* ≥2 nights per month awakened with nighttime symptoms
* Some limitation of activity
* ≥2 episodes of asthma during the past year that have required systemic corticosteroids.

Exclusion Criteria:

* Significant underlying respiratory disease other than asthma (such as cystic fibrosis or chronic lung disease) that could potentially interfere with asthma-related outcome measures.
* Significant co-morbid conditions (such as moderate to severe developmental delay, i.e. special education classroom or diagnosis) that could preclude participation in an education-based intervention.
* Inability to speak or understand English (child or parent).
* Children in foster care or other situations in which consent cannot be obtained from a guardian.
* Prior enrollment in the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Moorman JE, Rudd RA, Johnson CA, King M, Minor P, Bailey C, Scalia MR, Akinbami LJ; Centers for Disease Control and Prevention (CDC). National surveillance for asthma--United States, 1980-2004. MMWR Surveill Summ. 2007 Oct 19;56(8):1-54. PMID 17947969
- [Background] Akinbami LJ, Moorman JE, Garbe PL, Sondik EJ. Status of childhood asthma in the United States, 1980-2007. Pediatrics. 2009 Mar;123 Suppl 3:S131-45. doi: 10.1542/peds.2008-2233C. PMID 19221156
- [Background] Forero R, Bauman A, Young L, Larkin P. Asthma prevalence and management in Australian adolescents: results from three community surveys. J Adolesc Health. 1992 Dec;13(8):707-12. doi: 10.1016/1054-139x(92)90068-m. PMID 1290773
- [Background] Kyngas HA. Compliance of adolescents with asthma. Nurs Health Sci. 1999 Sep;1(3):195-202. doi: 10.1046/j.1442-2018.1999.00025.x. PMID 10894643
- [Background] Braun-Fahrlander C, Gassner M, Grize L, Minder CE, Varonier HS, Vuille JC, Wuthrich B, Sennhauser FH. Comparison of responses to an asthma symptom questionnaire (ISAAC core questions) completed by adolescents and their parents. SCARPOL-Team. Swiss Study on Childhood Allergy and Respiratory Symptoms with respect to Air Pollution. Pediatr Pulmonol. 1998 Mar;25(3):159-66. doi: 10.1002/(sici)1099-0496(199803)25:33.0.co;2-h. PMID 9556007
- [Background] Venn A, Lewis S, Cooper M, Hill J, Britton J. Questionnaire study of effect of sex and age on the prevalence of wheeze and asthma in adolescence. BMJ. 1998 Jun 27;316(7149):1945-6. doi: 10.1136/bmj.316.7149.1945. No abstract available. PMID 9641931
- [Background] National asthma education and prevention program expert panel report 3: Guidelines for the Diagnosis and Management of Asthma. National Heart Lunch and Blood Institute. 2007:NIH Publication No. 07-4051.
- [Background] Anhoj J, Moldrup C. Feasibility of collecting diary data from asthma patients through mobile phones and SMS (short message service): response rate analysis and focus group evaluation from a pilot study. J Med Internet Res. 2004 Dec 2;6(4):e42. doi: 10.2196/jmir.6.4.e42. PMID 15631966
- [Background] Nathan RA, Sorkness CA, Kosinski M, Schatz M, Li JT, Marcus P, Murray JJ, Pendergraft TB. Development of the asthma control test: a survey for assessing asthma control. J Allergy Clin Immunol. 2004 Jan;113(1):59-65. doi: 10.1016/j.jaci.2003.09.008. PMID 14713908
- [Background] Mosnaim GS, Cohen MS, Rhoads CH, Rittner SS, Powell LH. Use of MP3 players to increase asthma knowledge in inner-city African-American adolescents. Int J Behav Med. 2008;15(4):341-6. doi: 10.1080/10705500802365656. PMID 19005935

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile-based Asthma Action Plan: The mobile phone based application features will include ambulatory peak flow and asthma symptoms diary, individualized treatment plan for routine care and during episodes of acute asthma symptoms, and education components to reinforce asthma self-management concepts.
  Mobile-based Asthma Action Plan : The participant will be distributed a mobile phone (iPhone or Android) at the time of consent. The mobile-based Asthma Action Plan application will be provided on the mobile device. The mobile phone based application features will include ambulatory peak flow and asthma symptoms diary, individualized treatment plan for routine care and during episodes of acute asthma symptoms, and education components to reinforce asthma self-management concepts. Participants will receive 3 daily messages from the Asthma Action Plan mobile application. A fourth "rotating" message will be sent twice weekly.
Period: Overall Study
Arm/Group | Mobile-based Asthma Action Plan
Started | 22
Completed | 20
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mobile-based Asthma Action Plan
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Mobile Asthma Action Plan (AAP) Usage
Description: Median number of days per week (range 0-7) the Asthma Action Plan was utilized to record routine (daily) symptoms or peak flow measurements.
Time Frame: Eight weeks
Measure: Median (Full Range); unit: days per week
Arm/Group | Mobile-based Asthma Action Plan
Number analyzed (Participants) | 20
days per week | 4.3 [0 to 7]

2. Secondary Outcome: Number of Participants That Utilized the Asthma Action Plan
Description: The frequency of utilization of the Asthma Action Plan for acute symptoms among the study population will be measured and compared to responses of daily prompts that will ask participants to record whether they used rescue medication.
Time Frame: Eight weeks
Measure: Number; unit: participants
Arm/Group | Mobile-based Asthma Action Plan
Number analyzed (Participants) | 20
participants | 11

3. Secondary Outcome: Asthma Self-Efficacy for Adolescent Children
Description: The Child Self-Efficacy instrument is a 14 item validated questionnaire designed to measure the child's self-efficacy with regard to attack prevention and attack management. The child will be required to select one of 5 responses ranging from "not at all sure" (1 point); "a little bit sure" (2 points); "fairly sure" (3 points); "quite sure" (4 points) to "completely sure" (5 points). Total score range from 14-70. The higher score represent a greater degree of self-efficacy. The Cronbach's α reliability = 0.75. The child self-efficacy questionnaire will be administered at baseline (pre-intervention) and at the end of the intervention (post-intervention).
Time Frame: Baseline and eight weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile-based Asthma Action Plan
Number analyzed (Participants) | 20
units on a scale
  Eight Weeks (Post-Intervention) | 62.8 (5.7)
  Baseline | 57.2 (9.1)

4. Secondary Outcome: Asthma Control Test™ Scores
Description: The Asthma Control Test™ (ACT) is a 5 question health survey used to measure asthma control in individuals 12 years of age and older. The total sum scores range from 5-25. Higher scores mean that asthma is more controlled. The ACT is an efficient, reliable, and valid method of measuring asthma control, with or without, lung functioning measures such as spirometry. ACT helps identify and detect asthma patients who are not well controlled. ACT scores were examined pre- and post-intervention. A score total of 19 or less means asthma may not be well controlled. The timeframe is during the past 4 weeks. The scale range for Question 1 is "all the time" (1) to "none of the time" (5); Question 2 range: "more than once a day" (1) to "not at all" (5); Question 3 range: "4 or more nights a week" (1) to "not at all" (5); Question 4 range: "3 or more times per day" (1) to "not at all" (5); Question 5 range: "not controlled at all" (1) to "completely controlled" (5).
Time Frame: Baseline and eight weeks
Population: All participants and participants with uncontrolled asthma at baseline. The number of participant with uncontrolled asthma 10.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile-based Asthma Action Plan
Number analyzed (Participants) | 20
units on a scale
  Eight Weeks, All Participants | 20.3 (3.94)
  Baseline All Participants | 19.4 (4.63)
  Participants with Uncontrolled Asthma, Baseline | 15.3 (2.5)
  Participants with Uncontrolled Asthma, Eight Weeks | 19.1 (4.2)
Statistical Analysis 1: Comparison: Mobile-based Asthma Action Plan; This a comparison for participants with uncontrolled asthma at baseline and change in scores over time; Test type: Superiority or Other; p = 0.03, ANCOVA

ADVERSE EVENTS:
Description: There were zero adverse events that occurred.
Arm/Group | Mobile-based Asthma Action Plan
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
There are no limitations/caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes